CLINICAL TRIAL: NCT06145061
Title: Evaluation on Biological Characteristics of Acupoints in Premature Ovarian Insufficiency:A Case-control Study Protocol.
Brief Title: Evaluation on Biological Characteristics of Acupoints in Premature Ovarian Insufficiency
Status: Recruiting | Type: Observational
Sponsor: Xiaomei Shao (Other)
Responsible Party: Sponsor-Investigator, Xiaomei Shao, Professor, The Third Affiliated hospital of Zhejiang Chinese Medical University
Organization: The Third Affiliated hospital of Zhejiang Chinese Medical University (Other)
Other Study IDs: 2023ZX010-POI
Record Dates: First submitted 2023-11-18; First posted 2023-11-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Premature Ovarian Insufficiency
Keywords: Acupuncture; Biological Characteristics of Acupoint Representation; infrared thermal imaging; pain threshold testing
MeSH Terms: conditions — Primary Ovarian Insufficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- POI patients: POI patients:1.meet the diagnostic criteria for POI:POI diagnostic criteria refer to the 2016 European Society for Reproductive Medicine POI guidelines:Age < 40 years; Oligomenorrhea or amenorrhea for at least 4 months; Two measurements (on day 2-4 of the menstrual cycle, at least 4 weeks apart)Follicle Stimulating Hormone（FSH） > 25 IU/L and meet the above three requirements.2.18 years old ≤ age < 40 years old, gender female; 3.They are conscious and able to communicate normally.4.Provide recent transvaginal ultrasound or pelvic color Doppler ultrasound examination report to determine the menstrual cycle.5.Those who understand and are willing to comply with the study protocol and sign the informed consent form.
  Interventions: Device: all patients and healthy people will receive at least 3 infrared thermal imaging examinations of acupoints and pain threshold examinations of acupoints.
- healthy subjects: Healthy subjects:1.Healthy subjects who can provide physical examination report within the past 1 year and have routine physical examination by the investigator, and confirm that they have no serious underlying diseases such as reproductive system, urinary system, blood, endocrine system and nervous system;2.Currently no symptoms of oligomenorrhea or amenorrhea;3.18 years ≤ age < 40 years, female;4.Those who understand and are willing to comply with the study protocol and sign the informed consent form.
  Interventions: Device: all patients and healthy people will receive at least 3 infrared thermal imaging examinations of acupoints and pain threshold examinations of acupoints.

INTERVENTIONS:
Device: all patients and healthy people will receive at least 3 infrared thermal imaging examinations of acupoints and pain threshold examinations of acupoints. — Infrared thermal imaging detection scheme of acupoints:Detection equipment NEC R550 infrared thermal imager.Records the corresponding acupoints coordinates,and starts to collect the infrared thermal image.and 6 images will be taken continuously for each detected part.The infrared thermograms were stored and extract the temperature values of the corresponding coordinates of the acupoints.The average temperature values of the acupoints in the six infrared thermograms were calculated as their temperatures.Pain threshold detection scheme of acupoints:The instrument and equipment use the FDX25 hand-held pain threshold test instrument to explore the acupoints.Place the probe of the pain measuring instrument vertically on the pain measuring acupoint, slowly and steadily press downward at a constant speed, and stop pressing immediately when the subject begins to feel pain. At this point, the reading on the display is the subject's pain threshold. All acupoints shall be measured once in total.

SUMMARY:
Acupuncture has been widely used in the treatment of Premature Ovarian Insufficiency(POI), but the selection of acupoints is indeterminate and lacks biological basis.In recent years,some studies suggested the "acupoint sensitization",that is,changes such as pain sensitivity and heat sensitivity appear on the acupoints under disease state.The biological characteristics of acupoints can reflect the state of local tissue and might be a potential factor for guiding acupoint selection. This study aims to compare the temperature and pain threshold of acupoints between POI patients and the healthy population.At the meantime,clinical diagnosis of POI is based on clinical symptoms and Follicle Stimulating Hormone (FSH).However,FSH fluctuates so much that prediction accuracy is not high and clinical application is limited.Therefore, given the lack of proper diagnostic accuracy in POI and the concept of "acupoint sensitization",it is necessary to summarize the changes of biological characteristics of related acupoints under physiological and pathological conditions as an auxiliary means to improve the diagnostic rate of POI.

DETAILED DESCRIPTION:
The study is a case-control study protocol involving 150 POI patients from three clinical centers and 150 healthy persons in China.The duration of the study is one year, and all patients and healthy people will receive at least 3 infrared thermal imaging examinations of acupoints and pain threshold examinations.The primary outcome is to investigate the difference in the skin temperature and pain threshold of acupoints between POI and healthy persons.In the meanwhile,we will collect FSH, serum estradiol (E2) and some relevant scales,including modified Kupperman Index,Zung's Self-Rating Anxiety Scale(SAS),Zung's Self-Rating Depression Scale(SDS),Traditional Chinese medicine(TCM) constitution scale as second outcomes.

ELIGIBILITY:
Inclusion Criteria:

- POI patient inclusion criteria:1.meet the diagnostic criteria for POI:POI diagnostic criteria refer to the 2016 European Society for Reproductive Medicine POI guidelines:Age < 40 years; Oligomenorrhea or amenorrhea for at least 4 months; Two measurements (on day 2-4 of the menstrual cycle, at least 4 weeks apart)Follicle Stimulating Hormone（FSH） > 25 IU/L and meet the above three requirements.

2.18 years old ≤ age < 40 years old, gender female; 3.They are conscious and able to communicate normally. 4.Provide recent transvaginal ultrasound or pelvic color Doppler ultrasound examination report to determine the menstrual cycle.

5.Those who understand and are willing to comply with the study protocol and sign the informed consent form.

Healthy volunteers inclusion criteria:1.Healthy subjects who can provide physical examination report within the past 1 year and have routine physical examination by the investigator, and confirm that they have no serious underlying diseases such as reproductive system, urinary system, blood, endocrine system and nervous system;2.Currently no symptoms of oligomenorrhea or amenorrhea;3.18 years ≤ age < 40 years, female;4.Those who understand and are willing to comply with the study protocol and sign the informed consent form.

Exclusion Criteria:

- POI patient exclusion criteria:Patients who met any of the following criteria were excluded:1.low response or no response to exogenous gonadotropin, congenital reproductive tract dysplasia;2.Subjects who are pregnant or lactating;3.Patients with abnormal body temperature were found before detection;4.patients with mental illness, severe depression, alcohol dependence, history of drug abuse or serious primary diseases such as cardiovascular, liver, kidney and hematopoietic system; 5.Patients who do not cooperate with the study protocol of this study

Healthy volunteers exclusion criteria:volunteers who met any of the following criteria were excluded:1.mentally ill patients, patients with severe depression, alcohol dependence or those with a history of drug abuse;2.Subjects who are pregnant or lactating;3.volunteers with abnormal body temperature before testing;4.Those who do not cooperate with the study protocol of this study

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Premature Ovarian Insufficiency refers to the clinical symptoms of ovarian dysfunction in women before the age of 40, mainly manifested as abnormal menstruation,elevated gonadotropin levels and fluctuating decline in estrogen levels.Currently,POI is diagnosed clinically in patients <40 years of age with abnormal menstruation (amenorrhea or oligomenorrhea>4 months) and FSH>25U/L (two consecutive measurements more than 4 weeks apart).However,FSH fluctuates so much that prediction accuracy is not high and clinical application is limited.The global incidence of POI is 1%,and it is about 2.8% in China.In the long run, POI patients face various health risks, such as increased incidence of cardiovascular diseases, bone and joint diseases, genitourinary diseases, psychological diseases,etc.,and may even lead to shortened life expectancy, which seriously endangers women's physical, psychological and social aspects.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
The difference in the temperature and pain threshold of acupoints between POI and healthy populations | Baseline,6 months after,12 months after.
  The primary objective of this study is to investigate the difference in the temperature and pain threshold of acupoints between POI and healthy populations.

SECONDARY OUTCOMES:
Modified Kupperman | Baseline,6 months after,12 months after.
  The modified Kupperman Index consists of 13 items . In addition to the same 11 items included in the original Index,the modified version adds urogenital symptoms, including urinary infection and sexual complaints. The original 11 items included sweating/hot flushes, palpitation, vertigo, headache, paresthesia, formication, arthralgia, and myalgia (categorized as somatic symptoms), and fatigue, nervousness, and melancholia categorized as psychological symptoms. A scale ranging from 0 to 3 points is used to describe the severity of the complaints. The weighting factors were the same as those used in the original KI, and provide two points for both urogenital symptoms. The total score ranges from 0 to 63, calculated as the sum of all items by the weighting factor. Scores ranging from 0-6, 7-15, 16-30, and >30 were used to rate the degree of severity as none, mild, moderate, and severe, respectively.
Zung's Self-Rating Anxiety Scale(SAS) | Baseline,6 months after,12 months after.
  The SAS is used to assess the subjective feelings of patients with anxiety. SAS has good psychometric credentials, and it is suitable for all types of psychiatric disorders in which anxiety symptoms are predominant. There are 20 items on a four-point scale, and higher scores indicate greater anxiety.SAS has good psychometric credentials and can assist in the assessment of patients' anxiety status.
Zung's Self-Rating Depression Scale(SDS) | Baseline,6 months after,12 months after.
  The SDS can reflect the depressive state and its variability well (Zung, 1965). The scale contains 20 items scored on a 4-point scale. The rough scores were obtained by summing each of the 20 new items, multiplying the rough scores by 1.25, and then taking the integer part as the standard score. A standard score of 50-59 is considered to be a mild depressive mood, a standard score of 60-69 is considered to be moderate depression, and a standard score of more than 70 is considered to be severe depression. Patients respond according to their situation in the past week.
Traditional Chinese medicine(TCM) constitution scale | Baseline,6 months after,12 months after.
  TCM constitution scale is Prepared by Professor Wang Qi of Beijing University of Chinese Medicine, in order to evaluate peoplr's TCM constitution.Constitution classification is the basis and core content of TCM constitution research, which is to extract the relevant laws from the complex constitution phenomenon and finally build the constitution classification system.There are 9 items and 66 small items in the TCM constitution scale, which are required to be filled in according to the real situation in the last year. The results of the scale include nine constitutions: mild constitution, qi deficiency constitution, qi depression constitution, yin deficiency constitution, yang deficiency constitution, blood stasis constitution, special constitution, phlegm-dampness constitution and damp-heat constitution.
Follicle Stimulating Hormone | Baseline,6 months after,12 months after.
  Clinical diagnosis of POI is based on clinical symptoms and Follicle Stimulating Hormone (FSH).However,FSH fluctuates so much that prediction accuracy is not high and clinical application is limited

CONTACTS AND LOCATIONS:
Overall Officials: Xiaomei Shao, Ph.D, Principal Investigator — The Third Affiliated hospital of Zhejiang Chinese Medical University
Locations (1):
- the Third affiliated hospital of Zhejiang Chinese Medical university, Hangzhou, Zhejiang, China